CLINICAL TRIAL: NCT02154451
Title: Transient Infrared Imaging for Early Detection of Skin Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Skinfrared LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: 10-304
Record Dates: First submitted 2014-05-20; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Infrared Imaging Device- ALIAS — Infrared Camera

SUMMARY:
The hypothesis or study goal is to determine whether functional dynamic infrared imaging can be used for melanoma and other skin cancer screening and/or diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* All lesion in easily accessible places
* Lesion less than 3.5 cm

Exclusion Criteria:

* Any minors
* Lesion close to vital organs

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To detect skin cancers with >90% sensitivity and >50% specificity using infrared imaging | 5 years
  We are developing a screening algorithm than can compute data from infrared pictures and give us a threshold below which all the cases are benign and above which is malignant.
  Our primary outcome is to detect all the malignant cases with more than 90% sensitivity and all the benign cases with more than 50% specificity,

CONTACTS AND LOCATIONS:
Overall Officials: Sanchita krishna, PhD, Principal Investigator — Skinfrared LLC
Locations (3):
- United States (3):
  - University of New Mexico, Derm Clinic, Albuquerque, New Mexico
  - Univesity of New Mexico, Derm Clinic, Albuquerque, New Mexico
  - University of new Mexico, Dermatology clinic, Albuquerque, New Mexico